CLINICAL TRIAL: NCT01765569
Title: A Phase I, Open-Label, Multicenter, 3-Period, Fixed-Sequence Study To Investigate The Effect Of Vemurafenib On The Pharmacokinetics Of A Single Dose Of Digoxin In Patients With BRAFV600 Mutation-Positive Metastatic Malignancy
Brief Title: A Pharmacokinetics Study to Investigate the Effect of Vemurafenib on Digoxin in Patients With BRAFV600 Mutation-Positive Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO28394; 2012-003459-13 (EudraCT Number)
Record Dates: First submitted 2013-01-09; First posted 2013-01-10 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-08

CONDITIONS: Malignant Melanoma, Neoplasms
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — Digoxin; Vemurafenib

ARMS (1):
- Vemurafenib + Digoxin (Experimental): Single oral dose of digoxin 0.25 mg tablet on Day 1 in Period A, followed by vemurafenib 960 mg tablet orally BID from Day 8 to Day 28 in Period B, and then single oral dose of digoxin 0.25 mg on Day 29, and vemurafenib 960 mg orally BID from Day 29 to Day 35 in Period C.
  Interventions: Drug: Digoxin; Drug: Vemurafenib

INTERVENTIONS:
Drug: Digoxin — Participants received single oral dose of digoxin 0.25 mg tablet on Day 1 and Day 29.
Drug: Vemurafenib — Participants received vemurafenib 960 mg tablet orally BID from Day 8 to Day 35.

SUMMARY:
This open-label, multi-center, three-period, one sequence study will investigate the effect of vemurafenib on the pharmacokinetics of digoxin in patients with unresectable BRAFV600-mutation positive metastatic melanoma or other malignant tumor type that harbors a V600-activating mutation of BRAF without acceptable standard treatment options. Patients will receive multiple doses of vemurafenib in Periods B and C and a single dose of digoxin in Periods A and C. Eligible patients will have the option to continue treatment with vemurafenib as part of an extension study (NCT01739764). The anticipated time on study treatment is approximately 36 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients >= 18 years old
* Patients with either unresectable Stage IIIc or Stage IV metastatic melanoma positive for the BRAFV600 mutation or other malignant tumor type that harbors a V600-activating mutation of BRAF, as determined by results of cobas® 4800 BRAF V600 mutation test or a DNA sequencing method, and who have no acceptable standard treatment options
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Life expectancy >= 12 weeks
* Full recovery from the effects of any major surgery or significant traumatic injury within 14 days prior to the first dose of study treatment
* Adequate hematologic and end organ function
* Female patients of childbearing potential and male patients with partners of childbearing potential must agree to always use two effective methods of contraception
* Negative serum pregnancy test within 7 days prior to commencement of dosing in women of childbearing potential

Exclusion Criteria:

* Prior treatment with vemurafenib or other BRAF inhibitor within 42 days of first dose of study drug
* Prior anti-cancer therapy within 28 days before the first dose of study drug
* History of clinically significant cardiac or pulmonary dysfunction
* History of symptomatic congestive heart failure of any New York Heart Association class or serious cardiac arrhythmia requiring treatment
* History of myocardial infarction within 6 months prior to first dose of study drug
* Current dyspnea at rest, owing to complications of advanced malignancy or any requirement for supplemental oxygen to perform activities of daily living
* History of congenital long QT syndrome or QTc > 450 ms
* Current digoxin therapy or anticipated requirement to take digoxin therapy during the study
* Active central nervous system lesions
* Uncontrolled or poorly controlled diabetes
* Current severe, uncontrolled systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- Belarus (3):
  - Minsk
  - Minsk District
  - Vitebsk
- Israel (3):
  - Haifa
  - Tel Aviv
  - Tel Litwinsky
- Russia (3):
  - Kazan'
  - Moscow
  - Saint Petersburg
- Johannesburg, South Africa
- South Korea (2):
  - Daegu
  - Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- Vemurafenib + Digoxin: Single oral dose of digoxin 0.25 mg tablet on Day 1 in Period A, followed by vemurafenib 960 mg orally BID from Day 8 to Day 28 in Period B, and then single oral dose of digoxin 0.25 mg on Day 29, and vemurafenib 960 mg orally BID from Day 29 to Day 35 in Period C.
  Digoxin: Participants received single oral dose of digoxin 0.25 mg tablet on Day 1 and Day 29.
  Vemurafenib: Participants received vemurafenib 960 mg tablet orally BID from Day 8 to Day 35.
Period: Period A
Arm/Group | Vemurafenib + Digoxin
Started | 29
Completed | 29
Not Completed | 0
Period: Period B
Arm/Group | Vemurafenib + Digoxin
Started | 29
Completed | 28
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Period C
Arm/Group | Vemurafenib + Digoxin
Started | 28
Completed | 27
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vemurafenib + Digoxin
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUClast) of Digoxin
Description: AUClast = Area under the plasma-concentration time curve from time zero to the last measurable plasma concentration which is presented in hour*nanogram per milliliter (hour*ng/mL). Hour 0 (H0) signified pre-dose sampling.
Time Frame: Hour [H] 0, 0.5, 1, 2, 3, 4, 6, 8, 10-12 (Day [D] 1), 24, 30-32 (D2), 48 (D3), 72 (D4), 96 (D5), 168 (D8) post-digoxin dose; H0, 0.5, 1, 2, 3, 4, 6, 8, and 10-12H (D29), 24, 30-32 (D30), 48 (D31), 72 (D32), 96 (D33), 168 (D36) post digoxin dose
Population: PK Population included participants for whom PK data were collected.
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Groups:
- Period A (Digoxin): Participants received single oral dose of digoxin 0.25 mg tablet on Day 1.
- Period C (Digoxin + Vemurafenib): Participants received single oral dose of digoxin 0.25 mg tablet on Day 29 and vemurafenib 960 mg tablet orally BID from Day 29 to Day 35.
Arm/Group | Period A (Digoxin) | Period C (Digoxin + Vemurafenib)
Number analyzed (Participants) | 26 | 26
hour*ng/mL | 14.9 (4.22) | 27.7 (10.6)
Statistical Analysis 1: Comparison: Period A (Digoxin) vs Period C (Digoxin + Vemurafenib); Test type: Superiority or Other; Geometric Mean Ratio = 1.82, 90% CI 2-sided [1.63 to 2.02]

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUCinf) of Digoxin
Time Frame: as for outcome 1
Population: PK Population. Number of participants analysed = participants evaluable for the analysis.
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Period A (Digoxin) | Period C (Digoxin + Vemurafenib)
Number analyzed (Participants) | 11 | 11
hour*ng/mL | 18.5 (4.64) | 35.4 (4.16)

3. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC24) of Digoxin
Time Frame: as for outcome 1
Population: PK Population.
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Period A (Digoxin) | Period C (Digoxin + Vemurafenib)
Number analyzed (Participants) | 26 | 26
hour*ng/mL | 7.73 (1.86) | 10.6 (2.9)

4. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 168 Hours (AUC168) of Digoxin
Time Frame: as for outcome 1
Population: PK Population.
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Period A (Digoxin) | Period C (Digoxin + Vemurafenib)
Number analyzed (Participants) | 26 | 26
hour*ng/mL | 18.2 (4.85) | 29.7 (9.62)

5. Primary Outcome: Maximum Plasma Concentration (Cmax) of Digoxin
Time Frame: as for outcome 1
Population: PK Population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Period A (Digoxin) | Period C (Digoxin + Vemurafenib)
Number analyzed (Participants) | 26 | 26
ng/mL | 1.36 (0.408) | 1.99 (0.562)
Statistical Analysis 1: Comparison: Period A (Digoxin) vs Period C (Digoxin + Vemurafenib); Test type: Superiority or Other; Geometric Mean Ratio = 1.47, 90% CI 2-sided [1.3 to 1.65]

6. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of Digoxin
Time Frame: as for outcome 1
Population: PK Population.
Measure: Median (Full Range); unit: hours
Arm/Group | Period A (Digoxin) | Period C (Digoxin + Vemurafenib)
Number analyzed (Participants) | 26 | 26
hours | 1 [0.5 to 3] | 1 [0.47 to 2]

7. Primary Outcome: Terminal Half-Life (t1/2) of Digoxin
Time Frame: as for outcome 1
Population: PK Population. Number of participants analysed = participants evaluable for the analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Period A (Digoxin) | Period C (Digoxin + Vemurafenib)
Number analyzed (Participants) | 11 | 11
hours | 35 (8.67) | 56.4 (11)

8. Primary Outcome: Apparent Clearance (CL/F) of Digoxin
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population PK modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: as for outcome 1
Population: PK Population. Number of participants analysed = participants evaluable for the analysis.
Measure: Mean (Standard Deviation); unit: liters/hour
Arm/Group | Period A (Digoxin) | Period C (Digoxin + Vemurafenib)
Number analyzed (Participants) | 11 | 11
liters/hour | 14.5 (4.95) | 7.15 (0.808)

ADVERSE EVENTS:
Time Frame: From Screening to 28 days after the last dose of study treatment or until initiation of another anticancer therapy, whichever occurred first.
Groups:
- Period A: Single oral dose of digoxin 0.25 mg tablet on Day 1.
- Period B: Vemurafenib 960 mg orally BID from Day 8 to Day 28.
- Period C: Single oral dose of digoxin 0.25 mg on Day 29, and vemurafenib 960 mg orally BID from Day 29 to Day 35.
Arm/Group | Period A | Period B | Period C
Serious Adverse Events (participants affected / at risk) | 0/29 | 2/29 | 1/28
Other Adverse Events (participants affected / at risk) | 0/29 | 20/29 | 11/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period A (N=29) | Period B (N=29) | Period C (N=28)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period A (N=29) | Period B (N=29) | Period C (N=28)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 1 | 2
Asthenia (General disorders) | 0 | 1 | 4
Fatigue (General disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 7 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.